CLINICAL TRIAL: NCT04470258
Title: Elmo Respiratory Support Project for Patients With Hypoxemic Respiratory Insufficiency in Covid-19: Proof Of Concept and Usability
Brief Title: Elmo Respiratory Support Project - COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola de Saúde Pública do Ceará (Other Government)
Responsible Party: Principal Investigator, Marcelo Alcantara Holanda, Doctor, Escola de Saúde Pública do Ceará
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 4.104.233
Record Dates: First submitted 2020-06-10; First posted 2020-07-14 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: COVID-19; Respiratory Failure With Hypoxia
Keywords: COVID-19; Accute breathing failure; Continuous Positive Airway Pressure; Usability
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ELMO PROJECT AT COVID-19: PROOF OF CONCEPT AND USABILITY (Other): A realistic simulation will be carried out, centered on the heuristic evaluation, by a multiprofessional team (N= 6), to evaluate the performance of the new equipment in the execution of the pre-defined skills. The prototype will be tested on a mannequin by the research team and on healthy volunteers by health professionals, where physiological parameters and interface comfort will be evaluated.
  Interventions: Device: ELMO PROJECT AT COVID-19: PROOF OF CONCEPT AND USABILITY
- ELMO PROJECT AT COVID-19: STUDY IN HUMANS (Other): The second phase will consist of a clinical trial, in the application of the non-invasive respiratory device in 10 patients with respiratory failure by COVID-19, to assess its clinical effectiveness, through the analysis of the physiological variables and patient comfort.
  Interventions: Other: ELMO PROJECT AT COVID-19: STUDY IN HUMANS

INTERVENTIONS:
Other: ELMO PROJECT AT COVID-19: STUDY IN HUMANS — The Elmo system will be applied to 10 patients with hypoxemic respiratory failure by COVID-19 and its effectiveness will be assessed by analyzing the physiological variables and the patient's comfort, as well as their clinical outcomes (need for tracheal intubation) and recovery time. Hypoxemic respiratory failure and need for O2.
  Arms: ELMO PROJECT AT COVID-19: STUDY IN HUMANS
Device: ELMO PROJECT AT COVID-19: PROOF OF CONCEPT AND USABILITY — After testing for the following requirements: offering CPAP, ensuring the maintenance of alveolar ventilation without CO2 rebreathing, monitoring intra-ELMO pressure, minimizing adverse effects of the system such as noise, face temperature, airway dryness and comfort global; tests will be carried out on healthy volunteers using prototypes of the Elmo system and assessing whether their effectiveness in providing positive airway pressure and their usability from the perspective of their primary users (doctor, physiotherapist and nurses) and the volunteer's comfort . With this, realistic simulations will be carried out, centered on the evaluation based on heuristic principles.
  Arms: ELMO PROJECT AT COVID-19: PROOF OF CONCEPT AND USABILITY

SUMMARY:
The number of COVID-19 cases has been growing exponentially, so that the industrialized economies are facing a significant shortage in the number of ventilators available to meet the demands imposed by the disease. Noninvasive ventilatory support can be valuable for certain patients, avoiding tracheal intubation and its complications. However, non-invasive techniques have a high potential to generate aerosols during their implementation, especially when masks are used in which it is virtually impossible to completely prevent air leakage and the dispersion of aerosols with viral particles. In this context, a helmet-like interface system with complete sealing and respiratory isolation of the patient's head can allow the application of ventilatory support without intubation and with safety and comfort for healthcare professionals and patients. This type of device is not accessible in Brazil, nor is it available for immediate import, requiring the development of a national product. Meanwhile, a task force under the coordination of the School of Public Health (ESP) and Fundação Cearense de Apoio à Pesquisa (FUNCAP), with support from SENAI / FIEC and the Federal Universities of Ceará (UFC) and the University of Fortaleza (UNIFOR) advanced in the development of a prototype and accessory system capable of providing airway pressurization through a helmet-type interface, which was called the Elmo System.

DETAILED DESCRIPTION:
Objectives: 1. Validate the functionalities to fulfill the requirements and evaluate the usability of the Elmo System and 2. Evaluate the effectiveness of the Elmo system in the treatment of support to patients with hypoxemic respiratory failure caused by COVID-19.

Methods: This is a study divided into two stages. For objective 1, tests will be carried out on healthy volunteers using prototypes of the Elmo system and assessing whether their effectiveness in providing positive airway pressure and their usability from the perspective of their primary users (doctor, physiotherapist and nurses) and the comfort of the volunteer. After the tests to meet the requirements: continuous positive airway pressure (CPAP) offer, guarantee of the maintenance of alveolar ventilation without carbon dioxide (CO2) rebreathing, monitoring of intra-ELMO pressure, minimization of the adverse effects of the system such as noise, face temperature, dryness of the airways and overall comfort . In addition, realistic simulations will be carried out, centered on the assessment based on heuristic principles by a multiprofessional team with experience in mechanical ventilation, to assess the performance of the new equipment in the execution of the pre-defined skills. The second phase will consist of a clinical trial with application of the Elmo System to 10 patients with hypoxemic respiratory failure by COVID-19, to evaluate its effectiveness, through the analysis of physiological variables and patient comfort, as well as their clinical outcomes (need for tracheal intubation) and Insuf recovery time. Resp. Hypoxemic and need for O2 in a referral hospital for the treatment of this condition in Fortaleza / Ceara.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, age> or = 18 years, both sexes;
* Patient should be alert, oriented, and cooperative;
* When using oxygen therapy by CNO2> or = 4L/min, MR> or = 8 L/min of O2 or MV 50%, for maintain SpO2> 92%;
* Gasometric parameters (pre ELMO, up to 30 min before): pH> 7.35, PaO2> 60 mmHg;
* RX or chest CT scan with bilateral parenchymal opacities from the last 24 hours.

Exclusion Criteria:

* Exacerbation of Asthma, Chronic Obstructive Pulmonary Disease (COPD), pulmonary fibrosis or other lung diseases;
* Hemodynamic instability (SBP <90 mmHg or MBP <65 mmHg or need for vasoactive drugs);
* Pneumothorax or pneumomediastinum;
* Respiratory acidosis (pH <7.35 with PaCO2 >46mmHg);
* Signs of respiratory muscle fatigue (paradoxical breathing, accessory muscle use);
* Nausea or vomiting;
* Disorders of the auditory canal;
* Use of nasoenteric or nasogastric feeding tubes;
* Imminent risk of respiratory arrest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Usability tests of the Elmo system using Euristic usability principles | One week after all tests
  Usability test with the description of the identified problems of the main basic skills necessary for the correct handling of the non-invasive respiratory device (ELMO), through realistic simulations, severity scale and usability.
Evaluation of the effectiveness of the ELMO system using physiological parameters | One week after all tests
  To evaluate the effectiveness of the Elmo system in the supportive treatment of patients with hypoxemic respiratory failure caused by COVID-19 through peripheral oxygen saturation (%) before, during and after the application of Elmo.

SECONDARY OUTCOMES:
Evaluation of the effectiveness of the ELMO system using physiological parameters | One week after all tests
  To evaluate the effectiveness of the Elmo system in the supportive treatment of patients with hypoxemic respiratory failure caused by COVID-19 through respiratory rate (irpm) before, during and after the application of Elmo.
Evaluation of the effectiveness of the ELMO system using physiological parameters | One week after all tests
  To evaluate the effectiveness of the Elmo system in the supportive treatment of patients with hypoxemic respiratory failure caused by COVID-19 through heart rate before, during and after the application of Elmo.
Evaluation of the effectiveness of the ELMO system using physiological parameters | One week after all tests
  To evaluate the effectiveness of the Elmo system in the supportive treatment of patients with hypoxemic respiratory failure caused by COVID-19 through blood pressure before, during and after the application of Elmo.
Evaluation of the effectiveness of the ELMO system using physiological parameters | One week after all tests
  To evaluate the effectiveness of the Elmo system in the supportive treatment of patients with hypoxemic respiratory failure caused by COVID-19 through CO2 measurement at the end of exhalation (mmHg) before, during and after the application of Elmo.

CONTACTS AND LOCATIONS:
Overall Officials: MARCELO HOLANDA, Doctor, Principal Investigator — Escola de Saúde Pública do Ceará
Locations (1):
- Hospital Leonardo Da Vinci, Fortaleza, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tomaz BS, Gomes GC, Lino JA, Menezes DGA, Soares JB, Furtado V, Soares Junior L, Farias MDSQ, Lima DLN, Pereira EDB, Holanda MA. ELMO, a new helmet interface for CPAP to treat COVID-19-related acute hypoxemic respiratory failure outside the ICU: a feasibility study. J Bras Pneumol. 2022 Feb 2;48(1):e20210349. doi: 10.36416/1806-3756/e20210349. eCollection 2022. PMID 35137871